CLINICAL TRIAL: NCT05441033
Title: The Effects of Angel Sounds and Guided Imagery Technique Played to Expectant Couples on Attachment, Anxiety and Sleep Quality
Brief Title: The Effects of Angel Sounds and Guided Imagery Technique Played to Expectant Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Tuba Enise BENLI, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/2570
Record Dates: First submitted 2022-06-22; First posted 2022-07-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prenatal Anxiety; Prenatal Attachment; Sleep Quality
Keywords: Fetal Heart Rate Sounds; Guided Imagery; Prenatal Attachment; Anxiety, Pregnancy; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with three parallel arms: fetal heart sounds group (FHS), guided imagery technique group (GIT), and control group.
Masking Description: No masking was applied. Both participants and researchers were aware of the assigned interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-FHS (Experimental): Couples provided written and verbal consent after being informed about the study. Pre-test data were collected using the Personal Information Forms (PIF-Female, PIF-Male), Antenatal Mother Attachment Scale (PAAS), Antenatal Father Attachment Scale (PAAS), the Richard Campbell Sleep Questionnaire (RCSQ), and the State Anxiety Inventory (SAI).
  Couples listened to fetal heart sounds (angel sounds) each night before sleep for three consecutive nights, with each session lasting approximately 20 minutes. The researcher provided remote support via WhatsApp throughout the intervention period. Post-test data were collected on the fourth day using the same measurement tools.
  Interventions: Other: Fetal Heart Sounds (FHS) Listening Intervention
- Group-GIT (Experimental): Couples provided written and verbal consent after being informed about the study. Pre-test data were collected using the same tools as the FHS group. Couples were sent audio recordings prepared using guided imagery scripts, and instructed to listen each night before sleep for three consecutive nights. The audio included calming suggestions to promote attachment and reduce anxiety.
  On the fourth day, post-test data were collected using the same tools.
  Interventions: Other: Guided Imagery Technique (GIT) Intervention
- Control Group (No Intervention): Couples in the control group received no intervention. Pre-test data were collected using the same measurement tools as the experimental groups. After three days without intervention, post-test data were collected on the fourth day.

INTERVENTIONS:
Other: Fetal Heart Sounds (FHS) Listening Intervention — Pregnant women and their partners listened to fetal heart sounds (also referred to as angel sounds) for 20 minutes before bedtime on three consecutive nights using a fetal heart rate monitoring device. The intervention aimed to enhance prenatal attachment and reduce anxiety by increasing awareness of the fetus through auditory stimulation.
  Arms: Group-FHS
Other: Guided Imagery Technique (GIT) Intervention — Pregnant women and their partners listened to guided imagery audio recordings for 20 minutes before bedtime on three consecutive nights. The recordings were developed to support bonding with the baby, reduce anxiety, and improve sleep quality. The intervention was delivered via audio files prepared by the research team based on structured imagery scripts.
  Arms: Group-GIT

SUMMARY:
The study sample consisted of 177 pregnant women and their partners who met the inclusion criteria and participated in a prenatal education class. Expectant couples were randomized into three groups: Group 1 (FHS) listened to fetal heartbeat sounds, Group 2 (GIT) received the guided imagery intervention, and Group 3 served as the control group. Each group consisted of 59 couples.

DETAILED DESCRIPTION:
Aim: This randomized controlled trial aimed to evaluate the effects of listening to angel sounds (fetal heartbeat) and applying the guided imagery technique on prenatal attachment, anxiety, and sleep quality among expectant couples.

Methods: The study included 177 pregnant women and their partners who attended a prenatal education class and met the inclusion criteria. Expectant couples were randomly assigned into three equal groups. In Group 1 (FHS), only fetal heartbeat sounds were listened to. In Group 2 (GIT), the guided imagery technique was applied. Group 3 served as the control group. Each group consisted of 59 couples.

ELIGIBILITY:
Inclusion Criteria:

* Having basic literacy skills,
* Owning a smartphone and having internet access,
* Having a singleton and viable pregnancy,
* Being between the 27th and 38th weeks of gestation,
* Not having any diagnosed pregnancy-related risks (e.g., preeclampsia, diabetes, placenta previa, oligohydramnios),
* Not having any diagnosed fetal health issues (e.g., fetal anomalies, intrauterine growth restriction),
* Pregnant individuals and their spouses with no current or prior psychiatric diagnoses.

Exclusion Criteria:

* Not living with their spouse,
* Spouse working in shifts,
* Pregnancy via assisted reproductive techniques,
* Currently participating in childbirth education programs,
* Presence of communication difficulties or cognitive impairments in either the pregnant individual or the spouse.

Withdrawal Criteria:

* Participated in the intervention for fewer than 3 nights,
* Unable to use the Fetal Heart Rate Monitoring Device (FHRMD),
* Experiencing premature birth or pregnancy loss,
* Incomplete questionnaire data,
* Voluntary withdrawal from the study by the participant or their spouse. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
The Maternal Antenatal Attachment Scale | Change in Prenatal Attachment Levels of Expectant Mothers over 4 Days
  Each item of The Maternal Antenatal Attachment Scale (MAAS), which has a total of 19 items, focuses on the pregnant woman's feelings, attitudes and behaviors towards the fetus. The scale is likert-type and each item is scored between 1 and 5 (5=represents very strong feelings towards the fetus; 1=represents the absence of feelings towards the fetus). A high score indicates a high degree of attachment. 11 items in the scale are scored in the opposite direction (1, 3, 5, 6, 7, 9, 10, 12, 15, 16, 18).
The Paternal Antenatal Attachment Scale | Change in Prenatal Attachment Levels of Expectant Fathers over 4 Days
  The Paternal Antenatal Attachment Scale are based on the fathers' experiences in the last two weeks and measure the father's feelings and thoughts towards the developing fetus in the mother's womb. Increasing score indicates higher degree of attachment. The scale is in 5-point Likert type and consists of 16 items and two sub-dimensions. Sub dimensions; "quality of attachment [2, (3), (7), 9, 11, (12), (15), 16]" in which the emotional experience of the father is measured while thinking about the baby in the womb, "time spent on attachment [( 1), 4, (5), (6), (8), 10, (13), 14]". 9 items are reverse scored in the scale. Cronbach's alpha reliability coefficient of the scale was 0.82; the Cronbach's alpha of the quality of attachment sub-dimension was 0.80; The alpha of the time spent connecting sub-dimension is 0.67.
Richard Campbell Sleep Questionnaire | Change in Couples Sleep Quality over 4 Days
  This scale is a 6-item scale that measures the depth of night sleep, the time to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each of the items is evaluated on a chart with numbers from 0 to 100. According to the scale scoring, "0-25" points indicate very bad sleep, while "76-100" points indicate very good sleep. The 6th item, which evaluates the noise level in the environment, is excluded from the scale total score evaluation, and the total score is evaluated over 5 items. As the score of the scale increases, the sleep quality of the patients also increases. The scale's Cronbach α value is 0.91.
State Anxiety Inventory | Change in Couples State Anxiety over 4 Days
  The scale is a self-evaluation type scale consisting of short statements. It is used to determine how an individual feels in a certain situation and in a certain area. The emotions or behaviors expressed in the State Anxiety Scale items are answered by marking one of the options such as (1) not at all, (2) a little, (3) a lot, (4) completely, depending on the severity of the emotion or behavior. There are two types of expressions in the scale. These are reversed or straight forward expressions. reversed expressions; positive feelings express, direct expressions express negative feelings. When scoring reverse expressions, those with a weight of 1 are converted to 4, and those with a weight of 4 are converted to 1. In the State Anxiety Scale; There are ten reversed statements, items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. When scoring, the reversed and direct statements are summed.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Enise Benli, Phd, Principal Investigator — Giresun University
Locations (1):
- Faculty of Health Science, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers. The reason is that the institution where the study was conducted does not permit the distribution of individual-level data due to confidentiality policies.

REFERENCES:
- [Background] Benli TE, Aksoy Derya Y. Turkish validity and reliability study of Paternal Antenatal Attachment Scale. Perspect Psychiatr Care. 2021 Jan;57(1):295-303. doi: 10.1111/ppc.12563. Epub 2020 Jun 21. PMID 32567046
- See also: Related Info — https://bapsis.inonu.edu.tr/Default2.aspx